CLINICAL TRIAL: NCT00193661
Title: A Multi-Center, Open-Label, Observational Study of Testosterone Gel (1%) in the Treatment of Adolescent Boys With Hypogonadism
Brief Title: Observation Study of T-Gel (1%) in Treatment of Adolescent Boys With Hypogonadism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Solvay Pharmaceuticals (Industry)
Collaborators: Unimed Pharmaceuticals (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMD-01-090
Record Dates: First submitted 2005-09-11; First posted 2005-09-19 (Estimated); Last update posted 2015-01-16 (Estimated); Status verified 2006-09

CONDITIONS: Primary or Secondary Hypogonadism; Constitutional Delay in Growth and Puberty (CDGP)
Keywords: Hypogonadism
MeSH Terms: conditions — Hypogonadism

INTERVENTIONS:
Drug: Testosterone Gel (1%)

SUMMARY:
This study is to observe efficacy and safety after T-Gel 1% treatment in delayed puberty adolescents. Subjects who complete this trial may enter a 3 month extension study (UMD-01-090E).

ELIGIBILITY:
Inclusion Criteria:

* Primary or secondary hypogonadism or constitutional delay in growth and puberty (CDGP)

Exclusion Criteria:

* Skin intolerance to alcohol or allergy to soy
* Generalized skin disease
* Contraindication to testosterone or androgen products

Ages: 13 Years to 17 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2002-08; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Director Solvay, Study Director — Solvay Pharmaceuticals
Locations (19):
- United States (19):
  - Site 130, Birmingham, Alabama
  - Site 107, Los Angeles, California
  - Site 113, Sacramento, California
  - Site 114, Torrance, California
  - Site 121, Gainesville, Florida
  - Site 127, Jacksonville, Florida
  - Site 128, Jacksonville, Florida
  - Site 117, Indianapolis, Indiana
  - Site 111, Kansas City, Missouri
  - Site 129, Brooklyn, New York
  - Site 123, New York, New York
  - Site 131, Cincinnati, Ohio
  - Site 124, Columbus, Ohio
  - Site 103, Portland, Oregon
  - Site 109, Hershey, Pennsylvania
  - Site 125, Philadelphia, Pennsylvania
  - Site 126, Philadelphia, Pennsylvania
  - Site 104, Memphis, Tennessee
  - Site 205, Seattle, Washington